CLINICAL TRIAL: NCT03906812
Title: A Randomized Trial of Telemetry Compared With Unmonitored Floor Admissions in ED Patients With Low-Risk Chest Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of feasibility.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sean Collins, Sean Collins, M.D., MSc, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TeleVunmonitored
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Telemetry Usage; Chest Pain; Unstable Angina; Resource Utilization
MeSH Terms: conditions — Chest Pain; Angina, Unstable | interventions — Telemetry

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness - on admission, eligible, low-risk patients will be individually assigned to either unmonitored floor admission or floor admission with telemetry.
Who Masked: Outcomes Assessor
Masking Description: The study statistician will be blinded to study arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unmonitored floor admission (Active Comparator): Participants in this arm will be admitted to an unmonitored floor bed.
  Interventions: Other: Unmonitored
- Floor admission with telemetry (Active Comparator): Participants in this arm will be admitted to a telemetry bed.
  Interventions: Other: Telemetry

INTERVENTIONS:
Other: Telemetry — Bed type assignment
  Arms: Floor admission with telemetry
Other: Unmonitored — Bed type assignment
  Arms: Unmonitored floor admission

SUMMARY:
This study aims to determine, relative to telemetry admission, if admission to an unmonitored floor bed saves resources without an increased rate of adverse events in emergency department (ED) patients admitted with chest pain and low-risk features.

DETAILED DESCRIPTION:
Many patients admitted to the hospital with concern for cardiopulmonary and other acute illnesses are routinely placed on electrocardiographic monitoring (telemetry). Telemetry surveillance theoretically allows the clinical staff to monitor admitted patients for the development of both brady- and tachydysrhythmias. The goal is to identify dysrhythmias immediately via active cardiac monitoring in the very few patients who develop them, rather than identifying the dysrhythmia after the patient becomes symptomatic. However, the overwhelming majority (greater than 99 percent) of monitored patients do not experience any significant arrhythmia. The liberal use of monitoring in unnecessary situations may give the hospital staff a false sense of security and/or desensitize them to alarms. Studies also suggest the liberal use of telemetry inflates costs and clogs telemetry beds with little potential for benefit. These findings have contributed to the American Heart Association's statement that telemetry is of no benefit in patients with chest pain who are clinically low-risk or who are awake and alert and can describe their angina. Importantly, previous findings provide a foundation for identifying patients that do not need to undergo monitoring, but no study to date has rigorously prospectively applied these criteria in a randomized trial to determine the impact of selective telemetry utilization on clinical care and resources.

This study is a pragmatic, randomized, controlled trial of telemetry compared with unmonitored floor admissions in ED patients with low-risk chest pain. The primary aim is to determine, relative to telemetry admission, if admission to an unmonitored floor bed saves resources without an increased rate of adverse events in ED patients admitted with chest pain and low-risk features. In addition, the study will evaluate the effects of the same intervention in the same population on secondary outcomes including defibrillation, cardioversion or acute IV antiarrhythmic/vasoactive therapy. Finally, the study will associate reasons for telemetry exclusion, including provider discretion, with subsequent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patients admitted to the medical service at Vanderbilt University Medical Center with chest pain and low-risk clinical features.

Exclusion Criteria:

* Age less than 18 years
* Chest pain patients admitted to the ICU
* Patients with sickle cell disease
* Chest pain patients with high-risk electrocardiogram (ECG) criteria:
* abnormal but non-diagnostic of myocardial ischemia (prolonged PR, QRS, QTc intervals, new bundle branch blocks, left ventricular hypertrophy with strain)
* ischemia or prior infarction
* suggestive of acute myocardial infarction
* A positive troponin at any time during the current evaluation (above the 99 percent reference limit, greater than 0.03 nanograms per milliliter)
* Patients whom the admitting team feels has another non-low-risk indication for telemetry (e.g. acute heart failure, syncope with features concerning for a cardiac etiology, other arrhythmia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Total hospital resource utilization (costs) | ED to discharge (approximately 1 to 5 days)
  Total cost of the acute hospitalization and use of diagnostic testing and therapies

SECONDARY OUTCOMES:
Inhospital mortality | ED to discharge (approximately 1 to 5 days)
  Death in hospital - binary measurement
Total number of serious dysrhythmias by type | ED to discharge (approximately 1 to 5 days)
  Serious dysrhythmias resulting in defibrillation, cardioversion or acute intravenous (IV) antiarrhythmic/vasoactive therapy
Provider reasons for telemetry exclusion | ED to discharge (approximately 1 to 5 days)
  Association of reasons for telemetry exclusion, including provider discretion, with subsequent adverse events (e.g. death or serious dysrhythmias resulting in defibrillation, cardioversion or acute IV antiarrhythmic therapy)
Number of participants requiring transfer to the Intensive Care Unit (ICU) | ED to discharge (approximately 1 to 5 days)
  Measurement of whether or not a participant was transferred to the ICU
Total hospital and ED length of stay | ED to discharge (approximately 1 to 5 days)
  Total length of stay partitioned by location (ED, monitored bed, unmonitored bed etc.) measured in days
Rapid response team (RRT) call | ED to discharge (approximately 1 to 5 days)
  Dichotomous measure of whether or not the RRT was called and associated with arrhythmia or not
Cardiology consult | ED to discharge (approximately 1 to 5 days)
  Dichotomous measure of whether a cardiology consult was placed and associated with arrhythmia or not

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Collins, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Selker HP, Griffith JL, Dorey FJ, D'Agostino RB. How do physicians adapt when the coronary care unit is full? A prospective multicenter study. JAMA. 1987 Mar 6;257(9):1181-5. PMID 3806915
- [Background] Ward MJ, Eckman MH, Schauer DP, Raja AS, Collins S. Cost-effectiveness of telemetry for hospitalized patients with low-risk chest pain. Acad Emerg Med. 2011 Mar;18(3):279-86. doi: 10.1111/j.1553-2712.2011.01008.x. PMID 21401791
- [Background] Sandau KE, Funk M, Auerbach A, Barsness GW, Blum K, Cvach M, Lampert R, May JL, McDaniel GM, Perez MV, Sendelbach S, Sommargren CE, Wang PJ; American Heart Association Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; and Council on Cardiovascular Disease in the Young. Update to Practice Standards for Electrocardiographic Monitoring in Hospital Settings: A Scientific Statement From the American Heart Association. Circulation. 2017 Nov 7;136(19):e273-e344. doi: 10.1161/CIR.0000000000000527. Epub 2017 Oct 3. PMID 28974521
- [Background] Goldman L, Weinberg M, Weisberg M, Olshen R, Cook EF, Sargent RK, Lamas GA, Dennis C, Wilson C, Deckelbaum L, Fineberg H, Stiratelli R. A computer-derived protocol to aid in the diagnosis of emergency room patients with acute chest pain. N Engl J Med. 1982 Sep 2;307(10):588-96. doi: 10.1056/NEJM198209023071004. PMID 7110205
- [Background] Hollander JE, Valentine SM, McCuskey CF, Brogan GX Jr. Are monitored telemetry beds necessary for patients with nontraumatic chest pain and normal or nonspecific electrocardiograms? Am J Cardiol. 1997 Apr 15;79(8):1110-1. doi: 10.1016/s0002-9149(97)00057-x. PMID 9114775
- [Background] Snider A, Papaleo M, Beldner S, Park C, Katechis D, Galinkin D, Fein A. Is telemetry monitoring necessary in low-risk suspected acute chest pain syndromes? Chest. 2002 Aug;122(2):517-23. doi: 10.1378/chest.122.2.517. PMID 12171825
- [Background] Schull MJ, Redelmeier DA. Continuous electrocardiographic monitoring and cardiac arrest outcomes in 8,932 telemetry ward patients. Acad Emerg Med. 2000 Jun;7(6):647-52. doi: 10.1111/j.1553-2712.2000.tb02038.x. PMID 10905643
- [Background] Reaney PDW, Elliott HI, Noman A, Cooper JG. Risk stratifying chest pain patients in the emergency department using HEART, GRACE and TIMI scores, with a single contemporary troponin result, to predict major adverse cardiac events. Emerg Med J. 2018 Jul;35(7):420-427. doi: 10.1136/emermed-2017-207172. Epub 2018 Apr 5. PMID 29622596
- [Background] Estrada CA, Prasad NK, Rosman HS, Young MJ. Outcomes of patients hospitalized to a telemetry unit. Am J Cardiol. 1994 Aug 15;74(4):357-62. doi: 10.1016/0002-9149(94)90403-0. PMID 8059698
- [Background] Estrada CA, Rosman HS, Prasad NK, Battilana G, Alexander M, Held AC, Young MJ. Role of telemetry monitoring in the non-intensive care unit. Am J Cardiol. 1995 Nov 1;76(12):960-5. doi: 10.1016/s0002-9149(99)80270-7. PMID 7484840
- [Background] Hollander JE, Sites FD, Pollack CV Jr, Shofer FS. Lack of utility of telemetry monitoring for identification of cardiac death and life-threatening ventricular dysrhythmias in low-risk patients with chest pain. Ann Emerg Med. 2004 Jan;43(1):71-6. doi: 10.1016/s0196-0644(03)00719-4. PMID 14707944
- [Background] Lee TH, Juarez G, Cook EF, Weisberg MC, Rouan GW, Brand DA, Goldman L. Ruling out acute myocardial infarction. A prospective multicenter validation of a 12-hour strategy for patients at low risk. N Engl J Med. 1991 May 2;324(18):1239-46. doi: 10.1056/NEJM199105023241803. PMID 2014037